CLINICAL TRIAL: NCT03513666
Title: Toripalimab Combined With Pemetrexed Plus Carboplatin for Treatment of Recurrent or Advanced Non-small-cell Lung Cancer With EGFR-mutation Positive and T790M Negative After Progression on EGFR-TKI Treatment：a Multi-center, Single Arm Phase II Study
Brief Title: A Study of Toripalimab+ Pemetrexed Plus Carboplatin in Patients With EGFR-mutation Positive and T790M Negative After Progression on EGFR-TKI Treatment
Acronym: JS001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001-PII-LC-001
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): Toripalimab 240 mg or 360 mg Q3W in combination with chemotherapy
  Interventions: Combination Product: Drug intervention

INTERVENTIONS:
Combination Product: Drug intervention — anti-PD-1 monoclonal antibody Toripalimab injection combined with Pemetrexed and carboplatin

SUMMARY:
JS001 combined with pemetrexed plus carboplatin for treatment of recurrent or advanced non-small-cell lung cancer with EGFR-mutation positive and T790M negative after progression on EGFR-TKI treatment：a multi-center, single arm phase II study

ELIGIBILITY:
Inclusion Criteria:

Only the patients meeting all the following criteria can be eligible to participate in the trial:

* Histologically and/or cytologically confirmed advanced or recurrent non-small cell lung cancer with EGFR sensitive mutation (exon 19 deletion, exon 21 L858R), and meeting the following conditions at the same time:
* Previous first-line EGFR-TKI monotherapy with clinical benefit, followed by progression of disease;
* No exon 20 T790M mutation after failure of EGFR-TKI therapy;
* At least one measurable lesion (in accordance with RECIST 1.1);

Exclusion Criteria:

Patients who fulfill any of the following criteria must be excluded from the study:

* Histologically or cytopathologically confirmed combined with small cell lung cancer component or squamous cell carcinoma component >10%;
* Combined with other driver gene mutation with known drug therapy, including but not limited to ALK rearrangement, ROS1 mutation, BRAF600E mutation etc.;
* Previous systemic chemotherapy for advanced NSCLC;
* EGFR-TKI therapy within two weeks prior to enrollment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 12 weeks
  The primary endpoint is the antitumor activities in this study

SECONDARY OUTCOMES:
PFS | 18 months
  Progression free survival (PFS)
OS | 18 months
  Overall survival (OS)
DOR | 18 months
  Duration of response (DOR)

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Shanghai Pulmonary Hospita, Shanghai, Shanghai Municipality
  - Tangdu Hospital, Xi’an, Shanxi
  - The First Affiliated Hospital of Medical School of Zhejiang University, Hangzhou, Zhejiang
  - Zhengjiang Cancer Hospital, Hangzhou, Zhengjiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li LC, Chen XW, Fang L, Jian CL, Yu YX, Liao XY, Sun JG. YAP1 as a Novel Negative Biomarker of Immune Checkpoint Inhibitors for EGFR-Mutant Non-Small-Cell Lung Cancer. Can Respir J. 2023 Jun 21;2023:4689004. doi: 10.1155/2023/4689004. eCollection 2023. PMID 37388902